CLINICAL TRIAL: NCT04466800
Title: Functional and Respiratory Rehabilitation and Nutritional Care of COVID-19 Patients
Brief Title: Functional and Respiratory Rehabilitation and Nutritional Care of COVID-19 Patients (RECOVER-19)
Acronym: RECOVER-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC20_9875_RECOVER-19
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COVID
Keywords: COVID; Rehabilitation; Adapted physical activity; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, comparative, parallel-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group_rehabilitation program (Experimental): multidisciplinary and personalized rehabilitation program
  Interventions: Other: Intervention group_rehabilitation program
- Control group (No Intervention): Usual care of each site, including delivery of an information sheet concerning recommended physical activity (based on WHO recommendations) and nutrition. One month after inclusion, patients of this group will be offered a rehabilitation program (as described in the intervention group, but with only one session with a physical activity educator at home) and one dietitian consultation.

INTERVENTIONS:
Other: Intervention group_rehabilitation program — Regular physical activity, supervised by a physical education educator, a systematic malnutrition screening and a nutritional follow-up performed by a dietetician.
  Patients will follow a 4-week rehabilitation program, comprising 3 physical activity sessions per week for 4 weeks. First sessions will be supervised by a physical activity educator and patients will perform the following sessions at home, using physical training software. The physical activity educator will call patients once a week to ensure the sessions are correctly performed and adapt the program if necessary. Patients will also undergo a nutritional assessment carried out by a dietitian at the beginning of the program. A dietitian will call patients once a week to ensure their nutritional status is appropriate.
  Arms: Intervention group_rehabilitation program

SUMMARY:
Following the acute phase of COVID, some patients may have sequelae, such as breathing difficulties or malnutrition. We hypothesize that a functional and respiratory rehabilitation program associated with personalized nutritional care will improve quality of life, physical performance and respiratory capacities and will decrease the prevalence of malnutrition among those patients.

DETAILED DESCRIPTION:
In France, more than 150 000 patients have been infected by the SARS-CoV-2 virus and COVID has been responsible for more than 100 000 hospitalizations. Following the acute phase of this disease, some patients may have sequelae, such as breathing difficulties or malnutrition. However, the prevalence and intensity of those sequelae still remain unknown. Thus, a functional and respiratory rehabilitation program associated with personalized nutritional care may be necessary to improve those patients' prognosis.

This study aims to evaluate the effectiveness of a 4-week rehabilitation program following the acute phase of COVID. This program includes regular physical activity supervised by a physical acticity educator, a systematic malnutrition screening and a nutritional follow-up performed by a dietitian. Patients will be randomized in two groups: rehabilitation program (intervention group) or usual care (control group). Quality of life, physical performance, respiratory capacities and nutritional status will be assessed in both groups at inclusion and one month later (corresponding to the end of the rehabilitation program for the intervention group).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Laboratory (RT-PCR and/or serology) confirmed infection with SARS-CoV-2
* Date of first symptoms of SARS-CoV-2 infection > 4 weeks and < 4 months
* Persisting functional and/or respiratory deficit and/or asthenia and/or malnutrition beyond the first 4 weeks after COVID, defined as :
* Increase of mMRC (Modified Medical Research Council) score ≥ 1 between the month before COVID and beyond the first 4 weeks after COVID and/or
* Asthenia score (Pichot asthenia scale) > 22 beyond the first 4 weeks after COVID, if patient had no asthenia before COVID (asthenia score <8) and/or
* Weight loss > 5% within 6 months, comparing minimum weight between the month before COVID and beyond the first 4 weeks after COVID and/or
* BMI (Body Mass Index) < 20 (if age < 70 years) or < 22 (if age ≥ 70 years) if BMI (Body Mass Index) ≥ 20 (if age < 70 years) or ≥ 22 (if age ≥ 70 years) the month before COVID
* Patient affiliated to social security system
* Patient gave written informed consent

Exclusion Criteria:

* Patient unable to undergo a rehabilitation program due to comorbidities, such as major cardio-vascular disease or severe dementia
* Patient currently benefiting from physiotherapy sessions, in particular motor and / or respiratory therapy and / or an exercise re-training and / or respiratory rehabilitation program
* Patient living in a residential facility for dependent elderly people
* Patient not speaking french
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Impact of a multidisciplinary and personalized rehabilitation program on COVID patients's quality of life | 1 month
  Physical component score of the Short-Form 36 health survey between the beginning and the end of the rehabilitation program (from 0 to 100; highers scores mean better outcome)

SECONDARY OUTCOMES:
Impact of a multidisciplinary and personalized rehabilitation program in terms of Physical capacities | 1 month
  Number of repeated chair rises during 3 minutes
Impact of a multidisciplinary and personalized rehabilitation program in terms of Physical capacities | 1 month
  Aerobic physical capacity using Eval-DM software
Impact of a multidisciplinary and personalized rehabilitation program in terms of Respiratory capacities | 1 month
  Modified Medical Research Council scale (mMRC) (from 0 to 4, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Respiratory capacities | 3 months
  Modified Medical Research Council scale (mMRC) (from 0 to 4, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Respiratory capacities | 6 months
  Modified Medical Research Council scale (mMRC) (from 0 to 4, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Respiratory capacities | 1 month
  Borg scale (from 0 to 10, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Functional capacities | 1 month
  Barthel scale (from 0 to 100, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Functional capacities | 3 months
  Barthel scale (from 0 to 100, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Functional capacities | 6 months
  Barthel scale (from 0 to 100, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 1 month
  Weight loss
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 3 months
  Weight loss
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 6 months
  Weight loss
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 1 month
  Body mass index
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 3 months
  Body mass index
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 6 months
  Body mass index
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 1 month
  Muscular mass by brachial circumference or grip strength
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 1 month
  SEFI® score (from 0 to 10, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 3 months
  SEFI® score (from 0 to 10, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Malnutrition prevalence rate using GLIM malnutrition diagnostic criteria | 6 months
  SEFI® score (from 0 to 10, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of mortality | 1 month
  Mortality rate
Impact of a multidisciplinary and personalized rehabilitation program in terms of mortality | 3 months
  Mortality rate
Impact of a multidisciplinary and personalized rehabilitation program in terms of mortality | 6 months
  Mortality rate
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 1 month
  Score of the Short-Form 36 health Survey (from 0 to 100, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 3 months
  Score of the Short-Form 36 health Survey (from 0 to 100, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 6 months
  Score of the Short-Form 36 health Survey (from 0 to 100, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 1 month
  EuroQol 5 Dimensions 5 Levels surveys (from 0 to 1, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 3 months
  EuroQol 5 Dimensions 5 Levels surveys (from 0 to 1, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 6 months
  EuroQol 5 Dimensions 5 Levels surveys (from 0 to 1, highers scores mean better outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 1 month
  Proportion of patients returning to a professional activity
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 3 months
  Proportion of patients returning to a professional activity
Impact of a multidisciplinary and personalized rehabilitation program in terms of Quality of life | 6 months
  Proportion of patients returning to a professional activity
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 1 month
  Hospital and Anxiety Depression Scale (from 0 to 42, highers scores mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 3 months
  Hospital and Anxiety Depression Scale (from 0 to 42, highers scores mean worse outcome
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 6 months
  Hospital and Anxiety Depression Scale (from 0 to 42, highers scores mean worse outcome
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 1 month
  Pichot asthenia scale (from 0 to 32, highers mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 3 months
  Pichot asthenia scale (from 0 to 32, highers mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Anxiety and depression | 6 months
  Pichot asthenia scale (from 0 to 32, highers mean worse outcome)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 1 month
  Number of consultations with the healthcare professionals
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 3 months
  Number of consultations with the healthcare professionals
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 6 months
  Number of consultations with the healthcare professionals
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 1 month
  Rehospitalisation rate (all causes)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 3 months
  Rehospitalisation rate (all causes)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Healthcare consumption | 6 months
  Rehospitalisation rate (all causes)
Impact of a multidisciplinary and personalized rehabilitation program in terms of Medico-economic evaluation | 3 months
  Incremental cost-effectiveness ratio
Impact of a multidisciplinary and personalized rehabilitation program in terms of Medico-economic evaluation | 6 months
  Incremental cost-effectiveness ratio
Patient's opinion concerning the rehabilitation program | 3 months
  Satisfaction questionnaire with open-ended questions (no specific scale is available)
Patient's opinion concerning the rehabilitation program | 6 months
  Satisfaction questionnaire with open-ended questions (no specific scale is available)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Alix, Dr, Principal Investigator — Rennes University Hospital; Aranzazu PEDROSA GONZALEZ, Dr, Principal Investigator — Centre Hospitalier de Saint-Brieuc; Christophe POPINEAU, Dr, Principal Investigator — Centre Hospitalier Bretagne Atlantique; Patricia THOREUX, Pr, Principal Investigator — Hôtel Dieu Paris; Nadia SAIDANI, Dr, Principal Investigator — Centre Hospitalier de Cornouaille
Locations (5):
- France (5):
  - Hôtel Dieu Paris, Paris
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU Rennes, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - Centre Hospitalier Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No